CLINICAL TRIAL: NCT06202573
Title: The Effect of the Number of Steps on Edema and Ecchymosis Due to Rhinoplasty Surgery
Brief Title: Effect of Step Count on Edema After Rhinoplasty
Acronym: stepcount
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Salih Aydın, Prof.Dr., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: rhino-step
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Reduce Edema and Ecchymosis After Rhinoplasty
Keywords: Rhinoplasty; edeme; ecchymosis; step count
MeSH Terms: conditions — Ecchymosis | interventions — Rhinoplasty

STUDY DESIGN:
Intervention Model Description: prospective randomised self-controlled clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- group1A (Active Comparator): patients who have a step counter and we do not motivate them to walk
  Interventions: Procedure: rhinoplasty
- Group 1B (Active Comparator): patients who have a step counter, who do not motivate us to walk, and who will apply ice only on the 1st day after surgery
  Interventions: Procedure: rhinoplasty
- group 2 (Active Comparator): without step counter (only photos will be requested)
  Interventions: Procedure: rhinoplasty
- group 3 (Active Comparator): patients with step counters whom we motivate to take at least 5000 steps
  Interventions: Procedure: rhinoplasty
- group 4 (Active Comparator): patients with step counters whom we motivated to take at least 10000 steps
  Interventions: Procedure: rhinoplasty

INTERVENTIONS:
Procedure: rhinoplasty — patients who have a step counter and we do not motivate them to walk

SUMMARY:
Rhinoplasty surgery is being performed in increasing numbers in our country and around the world. After rhinoplasty surgery, patients experience swelling and bruising (ecchymosis) in their eyes. Many methods have been used to reduce this edema and bruising. Some of these methods are surgical techniques, medications, and supportive treatments used during and after surgery. (cortisol, vitamins, ice applications, etc.) When the literature is examined, there is currently no consensus on methods that reduce swelling and bruising. Again, in meta-analysis studies, there is no prominent or definitive method for reducing bruising and swelling. In our clinical observations, it has been observed that edema and bruising are significantly less common in tourists coming to our country from abroad. The idea that the reason for this may be that tourists walk a lot when they come to Istanbul, they want to travel a lot and see new places, has emerged as a hypothesis in our minds. The relationship between the number of steps taken during the day and postoperative edema-ecchymosis has not been examined before in the literature. In this respect, we think that our study will contribute to the literature.

DETAILED DESCRIPTION:
Edema and ecchymosis occurring in the eyes and face after rhinoplasty surgery greatly reduce the quality of life of patients. Many studies have been conducted in the literature to reduce this edema and ecchymosis. However, there is currently no successful method in the literature. Our aim in our study is to mobilize patients early after surgery and to investigate the effect of the number of steps they take after surgery on edema and attachment. For this purpose, 5 cohort groups will be created from patients who underwent rhinoplasty surgery by the same doctor. Patients will be randomly assigned to groups. The study was planned as a prospective, randomized, and self-controlled study.

Group 1A: patients who have a step counter and whom we do not motivate to walk Group 1B: patients who have a step counter, who do not motivate us to walk, and who will apply ice only on the 1st day after surgery Group 2: control group patients with and without step counters Group 3: patients who have a step counter and whom we motivate to take at least 5000 steps Group 4: patients with step counters, whom we motivated to take at least 10000 steps

Criteria for inclusion in the study: Having primary septorhinoplasty surgery under general anesthesia, being between the ages of 18-40, being the surgery patient of 3 researcher doctors (Dr. Salih Aydın, Dr. Timur Batmaz, Dr. Mehmet Erdil).

Criteria for inclusion in the study: revision septorhinoplasty surgery, patients with a chronic diagnosed disease such as diabetes, surgeries performed with conventional osteotomy, and surgeries without osteotomy. Measurements made with smartwatches other than the Xiaomi Band 5

The information of the patients participating in the study will be recorded on the forms. In this form: age, gender, accompanying diseases, smoking, drug use, occupation, doctor performing the surgery, duration of surgery (between intubation and extubation), end time of the surgery, the time he started walking on the first day, the number of steps taken on the first day and for 9 days. The daily step count (new day recordings will start at midnight) will be recorded. Patients will be asked to take facial photographs in the morning and evening. These photographs will be evaluated and noted using the edema-ecchymosis scale by a blind investigator. "Xiaomi Mi Band 5 smart bracelet" will be used to determine the number of steps taken. These wristbands will be given to the patients by the doctor performing the surgery and will be taken back at the end of the study. In light of the data obtained, the effect of early postoperative mobilization and the number of steps on edema and ecchymosis will be revealed.

ELIGIBILITY:
Inclusion Criteria:

* Having primary septorhinoplasty surgery under general anesthesia, being between the ages of 18-40, being the surgery patient of 3 research doctors (Dr. Salih Aydın, Dr. Timur Batmaz, Dr. Mehmet Erdil)

Exclusion Criteria:

* revision septorhinoplasty surgery, those with a chronic diagnosed disease such as concomitant diabetes, surgeries performed with conventional osteotomy, surgeries without osteotomy. Measurements made with smart watches other than Xiaomi band 5

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Step Count on Edema After Rhinoplasty | 6 months
  prospective study

CONTACTS AND LOCATIONS:
Overall Officials: Salih Aydin, Prof.Dr., Principal Investigator — İstinye Medical Faculty, Otorhinolaryngology department
Locations (1):
- Salih aydın, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No